CLINICAL TRIAL: NCT02720510
Title: A Randomized, Phase II Trial Evaluating the Efficacy and Safety of Lenalidomide, Bortezomib and Dexamethasone (RVD) With or Without Panobinostat in Transplant Eligible, Newly Diagnosed Multiple Myeloma
Brief Title: A Trial Evaluating Efficacy & Safety of RVD +/- Panobinostat in Transplant Eligible, Newly Diagnosed Multiple Myeloma (NDMM)
Acronym: PANORAMA4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A study was terminated due to low enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589DUS106
Record Dates: First submitted 2016-03-09; First posted 2016-03-28 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; farydak; panobinostat; LBH589; ASCT; transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - RVD + Pan (Active Comparator): Revlimid, Velcade, dexamethasone and Farydak
  Interventions: Drug: Revlimid; Drug: Velcade; Drug: dexamethasone; Drug: Farydak
- Arm 2 - RVD (Active Comparator): Revlimid, Velcade and Dexamethasone
  Interventions: Drug: Revlimid; Drug: Velcade; Drug: dexamethasone

INTERVENTIONS:
Drug: Revlimid — Revlimid was used with dexamethasone to treat patients with multiple myeloma
  Other Names: lenalidomide
Drug: Velcade — Velcade was a proteasome inhibitor indicated for treatment of patients with multiple myeloma
  Other Names: bortezomib
Drug: dexamethasone — Dexamethasone was a steroid used to treat patients with multiple myeloma.
  Other Names: Decadron
Drug: Farydak — FARYDAK® (panobinostat) capsules was a prescription medicine used, in combination with bortezomib and dexamethasone, to treat adults with a type of cancer called multiple myeloma after at least 2 other types of treatment have been tried.
  Other Names: panobinostat, LBH589
  Arms: Arm 1 - RVD + Pan

SUMMARY:
This was a multicenter, open-label, randomized phase II study which were to enroll 112 newly diagnosed symptomatic multiple myeloma patients in a 1:1 fashion. Patients were to enroll at approximately 20 centers in the United States.

Patients were to undergo stem cell mobilization with plerixafor plus Granulocyte Colony Stimulating Factor (G-CSF), according to investigator discretion, after 4 cycles of induction therapy. Study treatment interruption for stem cell collection were not to exceed 30 days. All patients were to receive one additional cycle of study treatment after stem cell collection and then proceed to autologous transplant using melphalan 200mg/m2(140mg/m2 for patients > 70 years), as conditioning.

After Autologus Stem Cell Transplant( ASCT), patients still on study were to initiate maintenance therapy within the 60-120 day period following ASCT, provided they have adequate blood count and clinical recovery. Patients in the RVD arm were to initiate maintenance therapy with lenalidomide alone, and patients in RVD-panobinostat arm were to receive lenalidomide + panobinostat maintenance. Lenalidomide were to be dosed orally at 10mg/day continuously in both arms, increasing to 15mg/day after the first 84 day cycle. Panobinostat were to be dosed at 10mg three times a week, every other week. Total planned duration of maintenance therapy were to be 3 years.

Patients were to remain on study treatment until they complete the maintenance phase, or until they experience disease progression, unacceptable toxicity, or at the discretion of the Investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient newly diagnosed with multiple myeloma, based on following IMWG 2014 definition (Rajkumar et al 2014):
* Clonal bone marrow plasma cells ≥ 10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events:
* Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder
* Any one or more of the following biomarkers of malignancy:

  1. Clonal bone marrow plasma cell percentage ≥ 60%
  2. Involved: uninvolved serum free light chain ratio ≥ 100
  3. >1 focal lesions on MRI studies
* Patient with measurable disease defined by at least 1 of the following conditions present at screening:
* Serum M-protein by Protein Electrophoresis (PEP) ≥ 1.0 g/dL (≥ 10 g/L).
* Urine M-protein by PEP ≥ 200 mg/24 hours. Involved serum free light chain level ≥ 10 mg/dL (≥ 100 mg/L), provided that the serum free light chain ratio is abnormal.
* Patient eligible for autologous stem cell transplantation based on the investigator's clinical judgment.
* Patient with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* Patient's age ≥ 18 and <75 years at time of signing the informed consent
* Patient provided written informed consent prior to any screening procedures
* Women of childbearing potential (WOCBP) with a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline

Key Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Any concomitant anti-cancer therapy (other than bortezomib/lenalidomide/dexamethasone; bisphosphonates are permitted only if commenced prior to the start of screening period)
* Unresolved diarrhea ≥ CTCAE grade 2 or presence of medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease).
* Allogeneic stem cell transplant recipient presenting with graft versus host disease either active or requiring immunosuppression
* Patient shown intolerance to bortezomib or to dexamethasone or components of these drugs or has any contraindication to one or the other drug, following locally applicable prescribing information
* Patient with rade ≥ 2 peripheral neuropathy or grade 1 peripheral neuropathy with pain on clinical examination at screening
* Patient received prior treatment with DAC inhibitors including Panobinostat
* Patient needing valproic acid for any medical condition during the study or within 5 days prior to first administration of panobinostat/study treatment.
* Patient taking any anti-cancer therapy concomitantly (bisphosphonates are permitted only if commenced prior to the start of screening period)
* Patient who received:

  1. prior anti-myeloma chemotherapy or medication including Immunomodulator (IMiDs) and Dex ≤ 3 weeks prior to start of study.
  2. experimental therapy or biologic immunotherapy including monoclonal antibodies ≤ 4 weeks prior to start of study.
  3. prior radiation therapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior start of study.
* Patient has not recovered from all therapy-related toxicities associated with above listed treatments to < grade 2 CTCAE.
* Patient undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy to < grade 2 CTCAE
* Patients with evidence of mucosal or internal bleeding
* Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 month prior to screening)
* Inability to determine the Fridericia's Correction Formula (QTc) F interval
* Patient with an impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g. ulcerative disease, uncontrolled nausea, vomiting, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
* Sexually active males unless they use a condom during intercourse while taking the drug during treatment, and for 6 months after stopping treatment
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - David Geffen School of Medicine at UCLA UCLA, Los Angeles, California
  - Memorial West Cancer Center Memorial Cancer Institute, Pembroke Pines, Florida
  - Northside Hospital Central Research Dept., Atlanta, Georgia
  - Oncology Hematology West Nebraska Cancer Specialists dbaNebraska Cancer Specialists, Omaha, Nebraska
  - Brooke Army Medical Center Hematology/Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 patients were randomized and treated in the study. None of the patient completed the study and all patients were discontinued.
Period: Overall Study
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Study Terminated by the sponsor | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (13.65) | 58.3 (3.51) | 60.5 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 2 | 1 | 3
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Near Complete Response (nCR)/CR Rate of the Combination of Panobinostat With Bortezomib, Lenalidomide and Dexamethasone (P-RVD) vs RVD in Newly Diagnosed Multiple Myeloma Patients
Time Frame: 84 days
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Minimal Residual Disease (MRD) Negativity (mCR) After 4 Cycles of Induction by Next Gen Sequencing
Description: MRD negativity by Clonal Sequencing (ClonoSEQTM) assay (Adaptive Biotechnologies)
Time Frame: Month 3
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Best Overall Response Rate (ORR) and MRD Negativity After ASCT and Maintenance
Description: ORR (CR + PR) and MRD negativity after ASCT and maintenance
Time Frame: Month 3 up to end of study, approximately 3 years.
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Depth of Response by International Myeloma Working Group (IMWG) Criteria
Description: Rate of Very Good Partial Response (VGPR), Complete Response (CR) and Stringent Complete Response (sCR)
Time Frame: Day 22 up to end of study, approximately 3 years
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response
Time Frame: From measurable response to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival
Time Frame: 3 years after the last patient is enrolled to the study
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated..
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Progression Free Survival
Time Frame: 3 years after the last patient is enrolled to the study
Population: The study was terminated prematurely and because only 6 patients were enrolled, efficacy data were not evaluated.
Arm/Group | Arm 1 - RVD + Pan | Arm 2 - RVD
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 1 year.
Groups:
- Arm 1- RVD+PAN: Revlimid, Velcade, dexamethasone and Farydak
Arm/Group | Arm 1- RVD+PAN | Arm 2 - RVD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- RVD+PAN (N=3) | Arm 2 - RVD (N=3)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- RVD+PAN (N=3) | Arm 2 - RVD (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated prematurely. The reason for study termination was not related to challenges linked to efficacy or safety data but instead, had faced unanticipated challenges with enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT02720510/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02720510/SAP_001.pdf